CLINICAL TRIAL: NCT06768892
Title: Workplace Weight Control Program: Combating Obesity in a Multinational Factory in Egypt.
Brief Title: Combating Obesity in a Workplace
Status: Not yet recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Noha Mohammed Elghazally, Assistant professor, Tanta University
Other Study IDs: obesity in a workplace
Record Dates: First submitted 2024-12-31; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Obesity | interventions — Diet Therapy; Cognitive Behavioral Therapy; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dietary Intervention — Each study participant will offer a tailored diet regimen according to age, sex, health status, physical activity and type of work either (office work or physical demanding work) after A 24-hour Dietary recall to calculate average calories requirements for each study participant separately. The participants' meals will be based on Mediterranean Diet and The Dietary Approaches to Stopping Hypertension (DASH Diet) as they proved effectiveness in lowering the risk of cardiovascular disease, insulin resistance, hypertension, obesity and Metabolic Syndrome. Dietary intervention aimed to the extent that 5-10% reduction in body weight, following the guideline of prevention and treatment of obesity.
  Other Names: Cognitive Behavioral Therapy (CBT); Physical exercise training
Behavioral: Cognitive Behavioral Therapy (CBT) — CBT method will be adapted and customized to facilitate a transition towards a heightened level of physical activity and to address the emotional and practical difficulties associated with weight loss. This encompassed assisting the participants in establishing attainable weight loss goals, identifying individualized approaches to manage appetite, sustaining healthy habits, and navigating social environments and circumstances related to food. The aforementioned factors were deliberated upon within the context of both group-based and individual settings, adhering to a meticulously customized guideline. This guideline encompassed the incorporation of positive thinking tactics, accompanied by assigned tasks to be completed between each session. The Cognitive Behavioral Therapy (CBT) intervention was administered as a 20-minute component within the weekly therapy sessions. cognitive-behavioral therapy (CBT) in conjunction with lif
Other: Physical exercise training — A weekly session of physical exercise training lasting 10 to 20 minutes will be incorporated at the workplace. The primary objective of the sessions was to increase muscle mass in the lower limbs for the purpose of sustaining physical capacity and boosting quiescent metabolism. The exercises comprised squats involving one or two legs, performed with or without dumbbells and core balls, as well as lunges performed while strolling forward and to each side. Additional exercises that emphasized overall strength encompassed shoulder and arm movements, as well as abdominal and back extension exercises. Participants were encouraged to execute the strength training exercises depicted in the program's takeout pamphlets twice per week. Furthermore, participants will be motivated to engage in aerobic leisure activities for a duration of two hours per week, including bicycling, walking, running, swimming, or participating in various sports.

SUMMARY:
Aim of the work: to assess the impact of 3-months workplace weight control program on both work ability and the severity of Metabolic Syndrome.

DETAILED DESCRIPTION:
Obesity is a significant public health concern worldwide. It is a multifactorial disease characterized by its complexity, as it is influenced by many factors as gut- brain axis, gut microbiome, genetics, behavioral, environmental ,and energy expenditure. A rising prevalence of obesity is observed in tandem with the acceleration of urbanization and economic transition.The obesity rate among employees and workers who constituting primarily the working population, has consequently witnessed a substantial surge and has garnered significant attention as a prominent public health issue.

According to (WHO), Egypt ranked 18th with highest prevalence of obesity globally and among the leading nations in obesity worldwide. The Prevalence of obesity among adults in Egypt in 2019 according to "100 million health survey" was 39.8% compared to 36% in 2017 in "STEP wise survey". In Egypt, the economic repercussions of obesity is nearly 62 Billion Egyptian pounds annually. This is the expense incurred for treatment comorbidities associated with obesity in adults which is direct health costs and indirect costs caused by decreased work abilities , work absenteeism, and may reach total disability.

Obesity is associated with metabolic abnormalities of metabolic syndrome (MetS). The prominent clinical features of this syndrome include abdominal adiposity, atherogenic dyslipidemia, the elevated blood pressure, insulin resistance, and proinflammatory and prothrombotic conditions.

The global prevalence of metabolic syndrome has been approximated to be approximately 25%. The observed rise in MetS is concomitant with the escalating prevalence of obesity. Obese populations have been associated with a greater prevalence of MetS, with values ranging from 59.6% to 75.7% of the individuals examined. According to the findings of the Centers for Disease Control and Prevention, there has been an observed rise in the prevalence of Metabolic Syndrome (MetS) among the adult population in the United States. Specifically, the prevalence has increased from 25.3% during the period of 1988-1994 to 34.2% during the period of 2007-2012. The subject of serious concern revolves around the impact of MetS within the working population, as it is closely linked to instances of job absenteeism resulting from illness, diminished productivity, and escalated healthcare expenditures.

Therefore, implementing of interventions aimed at preventing and treating MetS can significantly influence healthcare expenses and costs associated with short-term incapacity, while also enhancing job capacity. Emphasizing the potential for increased health-related productivity among the working population through the mitigation of metabolic syndrome severity.

The concept of work ability encompasses an individual's capacity to engage in work-related activities, and the intricate interplay between various cognitive, physical, and social factors, as well as the influence of diverse environmental elements. Obesity has a tremendous effect on the employee work ability, frequent absenteeism from work and long sick leave as obese workers and employees struggle to remain in the workforce.

Worksites are an appropriate setting and places of choice for implementing obesity intervention programs. An employee dedicates a significant amount of time to their work , and Workplaces possess various attributes, including well-established communication channels and social support systems, which have the potential to facilitate the implementation of multi-component, ecological, and individual interventions. In this context, the aim of our research is to implement 3- months obesity control program to improve work ability and to control the severity of the metabolic syndrome among of employees and workers in a multinational factory in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Manual workers and office employees
* BMI of ≥25 kg/m2 ,
* History of repeated sick leaves from work related health problems especially (musculoskeletal disorders (MSDs) and obesity related comorbidities as hypertension, diseases of the heart, hyperlipidemia ,Diabetes Mellitus and Metabolic syndrome)
* Age is above 18 years old

Exclusion Criteria:

* Age lower than 18
* BMI 24.9 and less

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: participants will involve manual workers and office employees who are manual workers and office employees who had BMI of ≥25 kg/m2 , history of repeated sick leaves from work related health problems especially musculoskeletal disorders (MSDs) and obesity related comorbidities as hypertension, diseases of the heart, hyperlipidemia ,diabetes and metabolic syndrome, and their age is above 18 years old .
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change of severity of the Metabolic Syndrome components | 3 months
  The change in the severity of the metabolic syndrome components following 3-months obesity control intervention in comparison with the baseline.
  All participants were assessed for the five criteria of metabolic syndrome (according to IDF&AHA): Metabolic syndrome was diagnosed if study Participants have at least three of the following five items: (1) Central obesity (waist circumference ≥ 102cm in male; ≥ 88 cm in female),(2) Blood pressure ≥130/85 mmhg,(3) Dyslipidemia (TG ≥ 150mg/dl), (4) Dyslipidemia (HDL-C < 40mg/dl in male; < 50mg/dl in female), and(5)Fasting blood glucose ≥ 110mg/dl.
  The blood pressure of participants in the office setting will be assessed and venous blood samples will be collected in order to assess blood lipids and fasting blood glucose levels. The safety blood profile will be conducted using established methodologies in a qualified laboratory specializing in clinical chemistry.

SECONDARY OUTCOMES:
Work Ability of participants | 3 months
  The Work ability of the study subjects will be measured before and after the obesity management intervention program using a standard questionnaire named Work Ability Index. The questionnaire comprises seven items, each utilizing a variable scoring system. The first assesses individual's present work capacity in relation to their best level of work capacity achieved in the past( 0 to 10). Second measures work capacity in respect to job expectations(2 to 10).Third pertains to the "number of current diseases diagnosed by a physician" (1to 7). The fourth pertains to the assessment of job impairment caused by diseases, (1 to 6). The fifth pertains to sick leave taken within the previous year, (1 to 5). sixth pertains to the individual's self-assessment of their work abilities during the past two years, (1, 4, or 7). Seventh element in the sequence is denoted as "mental resources" 1 to 4. WAI total score ranges from 2 to 49, low ( 2 - 27), medium (28 - 36), good(37-43),very good(44-49)

CONTACTS AND LOCATIONS:
Overall Officials: Rania El sallamy, Study Director — Tanta university faculty of medicine
Locations (1):
- Tanta University, Tanta, Egypt

REFERENCES:
- [Result] Andersen LL, Izquierdo M, Sundstrup E. Overweight and obesity are progressively associated with lower work ability in the general working population: cross-sectional study among 10,000 adults. Int Arch Occup Environ Health. 2017 Nov;90(8):779-787. doi: 10.1007/s00420-017-1240-0. Epub 2017 Jun 28. PMID 28660321
- [Result] Guzman M, Zbella E, Alvarez SS, Nguyen JL, Imperial E, Troncale FJ, Holub C, Mallhi AK, VanWyk S. Effect of an intensive lifestyle intervention on the prevalence of metabolic syndrome and its components among overweight and obese adults. J Public Health (Oxf). 2020 Nov 23;42(4):828-838. doi: 10.1093/pubmed/fdz170. PMID 31840755